CLINICAL TRIAL: NCT05361486
Title: Health Care Provider Use of Plasmodium Vivax Radical Cure (RC) With Tafenoquine or Primaquine After Semi-quantitative G6PD Testing: A Feasibility Study in Peru
Brief Title: Radical Cure (RC) With Tafenoquine or Primaquine After Semi-quantitative G6PD Testing: A Feasibility Study in Peru
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); UNITAID (Other); ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: MMV_TQ_21_01
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Malaria, Vivax
Keywords: Feasibility study, Tafenoquine, G6PD Testing
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Primaquine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Care Provider managing vivax patients in study facilities: All HCPs working in the selected facilities who are involved in the management of vivax patients will be approached to participate in the study.
  Interventions: Other: Training on revised algorithm; Other: Enhancing Pharmacovigilance; Other: Supervision of malaria services in selected facilities.
- Patients with confirmation of vivax, attending one of the study facilities: All patients aged 6 months onward, who have a confirmed P. vivax infection and who are in a study HF will be approached to participate in the study. This includes pregnant and lactating women, who have a contra-indication to both PQ and TQ, but for whom correct case management will be evaluated as part of the primary endpoints.
  Interventions: Diagnostic Test: G6PD testing; Drug: Tafenoquine; Drug: Primaquine; Other: Follow Up Visit at Day 3 [+2 days] after treatment start

INTERVENTIONS:
Other: Training on revised algorithm — relevant HCP working in study facilities will be trained on the relevant aspects of performing the G6PD testing, interpreting its result, evaluating patient's eligibility for RC and choosing the appropriate treatment as per their role accordingly
  Groups: Health Care Provider managing vivax patients in study facilities
Other: Enhancing Pharmacovigilance — Refresher training on PV reporting in the selected facilities. National PV forms will be reviewed and if required, modified in consultation with the national PV system.
  Groups: Health Care Provider managing vivax patients in study facilities
Other: Supervision of malaria services in selected facilities. — Supervisors in target regions will be trained as for the HCPs.
  Groups: Health Care Provider managing vivax patients in study facilities
Diagnostic Test: G6PD testing — G6PD test after Malaria Vivax diagnosis
  Groups: Patients with confirmation of vivax, attending one of the study facilities
Drug: Tafenoquine — 300 mg (2x150mg tablets) tafenoquine
  Other Names: Kozenis
  Groups: Patients with confirmation of vivax, attending one of the study facilities
Drug: Primaquine — 0.5mg/kg/7 days
  Groups: Patients with confirmation of vivax, attending one of the study facilities
Other: Follow Up Visit at Day 3 [+2 days] after treatment start — It will be checked if all patients have a Follow Up Visit at Day 3 [+2 days] after treatment start
  Groups: Patients with confirmation of vivax, attending one of the study facilities

SUMMARY:
The goal of this study is to evaluate the operational feasibility of using a new treatment algorithm for Malaria Vivax in Peru.

The implementation package includes the following interventions:

* A revised vivax treatment algorithm that incorporates new Radical Cure tools (G6PD test + Tafenoquine or Primaquine)
* The training of Health Care Providers ( HCPs) in the revised algorithm and the use of the new RC tools
* Patient counselling
* A follow-up visit at Day 3 [+2 days] for patients after treatment start
* Accompanying supporting measures: job aids, strengthening of supervision and PV processes

DETAILED DESCRIPTION:
The goal of this study is to evaluate the operational feasibility of providing Tafenoquine and Primaquine after semi-quantitative G6PD testing at different levels of the health services, in order to inform potential policy change, malaria strategy, and introduction planning.

This implementation research study will be carried out in Peru among 40 Health Care Providers ( HCPs) each treating a minimum of 15 patients with P. vivax malaria. The study will be conducted in Loreto Region (Loreto, Maynas and Ramon Castilla provinces), an area which is endemic for P. vivax.

A total of 30 health facilities will be included: 6 in the first phase and 12 will be added in the second phase. An additional 12 health facilities have been selected as backup in case the malaria case load is low, and this is needed in order to meet the sample size.

All relevant HCP working in study facilities will be trained on the relevant aspects of performing the G6PD testing, interpreting its result, evaluating patient's eligibility for Radical Cure and choosing the appropriate treatment as per their role accordingly.

HCP knowledge and skills regarding semi-quantitative G6PD testing and RC treatment will be assessed through standardized competency assessment (including self-assessments).

Adherence to the revised algorithm will be evaluated as follows. At each HF included in the study, the ideal patient case management cascade will be defined a priori. Individual HCP adherence to each step of the case management will be assessed against this cascade. By indexing each step in the patient care cascade to a specific HCP, the study will be able to consider feasibility at multiple levels, analysing adherence to specific steps of the case management algorithm.

A specific process will be put in place for patient counselling and standard tools such as a counselling checklist will be developed to assist HCPs. In addition, patient materials will be developed which will give explanations on the new Radical Cure tools, emphasize the need to come for a follow-up visit and outline the potential side effects that can be elicited by 8-AQ. Patients will be instructed to come back or call the facilities in case they experience those events.

The study will be carried out in following phases:

1. A formative research and baseline phase ( approx. 3 months) : this phase is meant to collect baseline information from the selected study facilities prior to introduction of the implementation package. This phase will also be important to field-test and validate study tools, such as the training material and documents and data collection tools (e.g. qualitative research questionnaires and interview guides). Finally, during this formative research phase, the supervision processes and tools will be revised.
2. A higher-level facilities phase ( approx. 8 months) : in this phase the implementation package will only be rolled out in selected higher-level facilities.

   An interim analysis will be conducted prior to rolling out the implementation package to lower-level facilities. The data cut-off point for this interim analysis will be once 50 patients have been treated with the revised algorithm. During this interim analysis, enrolment in Higher-level HF will continue.
3. An All-level facilities phase ( approx.14 months) : in this phase the implementation package will be rolled out to the lower-level facilities.

Final analysis will be performed at study end and results will be shared with the Peru National Malaria Control Program (NMCP) to make informed decisions on revisions to national malaria treatment policies.

The study aims to achieve the following specific objectives:

1. Assess HCP adherence to a revised case management algorithm for vivax malaria that involves providing RC treatment after semi-quantitative G6PD testing and a follow-up visit. This will be assessed at the provider, patient, and health facility (HF) level.
2. Determine the ability of HCP to safely implement RC treatment after semi-quantitative G6PD testing
3. Evaluate the quality and effectiveness of training and supervision strategies to support the implementation of semi-quantitative G6PD testing before RC treatment
4. Explore barriers and facilitators at the patient, provider, and facility level that mediate effective use of RC treatment with semi-quantitative G6PD testing. 5. Determine the costs associated with introducing semi-quantitative G6PD testing before RC treatment as part of routine care

ELIGIBILITY:
Inclusion Criteria Health Care Providers:

• All HCPs working in the selected facilities who are involved in the management of vivax patients.

Inclusion criteria patients:

* All patients aged 6 months onward, who have a confirmed P. vivax infection and who are treated in a study Health Facilities
* Pregnant and lactating women, who have a contra-indication to both Primaquine and Tafenoquine, but for whom correct case management will be evaluated as part of the primary endpoints.
* Patients providing informed consent and/or informed assent

Exclusion criteria patients:

• Patients with signs of severe infection

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * All Health Care Providers (HCPs) working in the selected facilities who are involved in the management of vivax patients
  * All patients aged 6 months onward, who have a confirmed P. vivax infection and who are treated in a Health Facility participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of HCP who adhere to the revised RC treatment algorithm as relevant to their role in patient case management. | Time from Malaria Vivax diagnosis until FU visit ( Day 3 [-1 day; +2 days]
  HCP will be assessed according to their roles such as performing the G6PD test, interpreting the test results, evaluating TQ/PQ ineligibility, prescribing treatment, administering treatment, and performing follow-up of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elmer Alejandro Llanos Cuentas, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia (UPCH)
Locations (1):
- Nauta Nucleo- Base, Nauta, Loreto, Peru

IPD SHARING:
Plan to Share IPD: Undecided
Considering to share study related information such as protocol, ICFs and final CSR after final publication has been published.

REFERENCES:
- [Background] Llanos-Cuentas A, Lacerda MV, Rueangweerayut R, Krudsood S, Gupta SK, Kochar SK, Arthur P, Chuenchom N, Mohrle JJ, Duparc S, Ugwuegbulam C, Kleim JP, Carter N, Green JA, Kellam L. Tafenoquine plus chloroquine for the treatment and relapse prevention of Plasmodium vivax malaria (DETECTIVE): a multicentre, double-blind, randomised, phase 2b dose-selection study. Lancet. 2014 Mar 22;383(9922):1049-58. doi: 10.1016/S0140-6736(13)62568-4. Epub 2013 Dec 19. PMID 24360369
- [Background] Anderle A, Bancone G, Domingo GJ, Gerth-Guyette E, Pal S, Satyagraha AW. Point-of-Care Testing for G6PD Deficiency: Opportunities for Screening. Int J Neonatal Screen. 2018;4(4):34. doi: 10.3390/ijns4040034. Epub 2018 Nov 19. PMID 31709308
- [Background] Chu CS, Bancone G, Kelley M, Advani N, Domingo GJ, Cutiongo-de la Paz EM, van der Merwe N, Cohen J, Gerth-Guyette E. Optimizing G6PD testing for Plasmodium vivax case management and beyond: why sex, counseling, and community engagement matter. Wellcome Open Res. 2020 Aug 25;5:21. doi: 10.12688/wellcomeopenres.15700.2. eCollection 2020. PMID 32766454
- [Background] Commons RJ, Simpson JA, Watson J, White NJ, Price RN. Estimating the Proportion of Plasmodium vivax Recurrences Caused by Relapse: A Systematic Review and Meta-Analysis. Am J Trop Med Hyg. 2020 Sep;103(3):1094-1099. doi: 10.4269/ajtmh.20-0186. PMID 32524950
- [Background] Domingo GJ, Advani N, Satyagraha AW, Sibley CH, Rowley E, Kalnoky M, Cohen J, Parker M, Kelley M. Addressing the gender-knowledge gap in glucose-6-phosphate dehydrogenase deficiency: challenges and opportunities. Int Health. 2019 Jan 1;11(1):7-14. doi: 10.1093/inthealth/ihy060. PMID 30184203
- [Background] Douglas NM, Poespoprodjo JR, Patriani D, Malloy MJ, Kenangalem E, Sugiarto P, Simpson JA, Soenarto Y, Anstey NM, Price RN. Unsupervised primaquine for the treatment of Plasmodium vivax malaria relapses in southern Papua: A hospital-based cohort study. PLoS Med. 2017 Aug 29;14(8):e1002379. doi: 10.1371/journal.pmed.1002379. eCollection 2017 Aug. PMID 28850568
- [Background] Edwards SJ, Braunholtz DA, Lilford RJ, Stevens AJ. Ethical issues in the design and conduct of cluster randomised controlled trials. BMJ. 1999 May 22;318(7195):1407-9. doi: 10.1136/bmj.318.7195.1407. No abstract available. PMID 10334756